CLINICAL TRIAL: NCT05668871
Title: Effects of Danning Tablet Under Lifestyle Intervention in Patients With Polypoid Lesions of Gallbladder: A Randomized, Open-labelled, Multicenter, Controlled Trial
Brief Title: A Study of Danning Tablet in Patients With Polypoid Lesions of Gallbladder
Acronym: PLG001
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Eastern Hepatobiliary Surgery Hospital (Other)
Responsible Party: Principal Investigator, Shen Feng, Professor and Chief Surgeon, Eastern Hepatobiliary Surgery Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CCPE202201
Record Dates: First submitted 2022-12-14; First posted 2022-12-30 (Actual); Last update posted 2022-12-30 (Actual); Status verified 2022-12

CONDITIONS: Polyps Gallbladder
Keywords: gallbladder; polyps; healthy lifestyle; herbal medicine; Danning Tablet
MeSH Terms: conditions — Polyps

STUDY DESIGN:
Intervention Model Description: Target population: Patients with multiple gallbladder polyps.
  Intervention and comparison:
  1. Test Group (N=168): Under lifestyle intervention, Danning Tablets will be taken orally 3 times each day, 5 tablets each time, from baseline to weeks 12±1.
  2. Controlled Group (N=168): Only in treatment of lifestyle intervention.
  Clinical Outcomes:
  1. Efficacy on shrinkage of gallbladder polyps and alleviation of clinical symptoms of gallbladder polyps.
  2. Safety in treatment of gallbladder polyps.
  Follow-up cycle: The length of follow-up cycle is 24 weeks, 5 visit windows (baseline, weeks 4±1, weeks 8±1, weeks 12±1, weeks 24±1) are set.
Masking Description: Open-labelled clinical trial, no masking involved.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Danning Tablet and lifestyle intervention group (Experimental): Under lifestyle intervention, Danning Tablet will be taken orally from baseline to weeks 12±1.
  Interventions: Drug: Danning Tablet
- Lifestyle intervention group (No Intervention): Lifestyle intervention only.

INTERVENTIONS:
Drug: Danning Tablet — 3 times each day, 5 tablets each time, take orally after meals.
  Other Names: Biliflow (NPN 80073325, manufactured by Shanghai Hutchison Pharmaceuticals Limited)
  Arms: Danning Tablet and lifestyle intervention group

SUMMARY:
The primary goal of this clinical trial is to evaluate the effect of Danning Tablet on shrinkage of gallbladder polyps compared to lifestyle intervention in 336 patients with gallbladder polyps. The main questions it aims to answer are:

* Medicine may be effective on shrinkage of gallbladder polyps and alleviation of clinical symptoms of gallbladder polyps.
* Chinese patent medicine (herbal medicine) may be safety in treatment of gallbladder polyps.

DETAILED DESCRIPTION:
Study design:

In this study, 336 participants will be randomly allocated to the test group or the controlled group in ratio of 1:1 and receive lifestyle intervention from baseline to weeks 24±1. However, in experimental group, participants will take Danning Tablet from baseline to weeks 12±1 (3 times each day, 5 tablets each time). In controlled group, only lifestyle intervention will be adopted. The length of follow-up cycle is 24 weeks.

Evaluation indicators:

Primary indicator: Changes in maximum diameter of gallbladder polyps, use gallbladder ultrasonography to evaluate this indicator on weeks 12±1 and weeks 24±1.

Secondly Indicators:

1. Changes in thickness of gallbladder wall, use gallbladder ultrasonography to evaluate this indicator on weeks 12±1 and weeks 24±1.
2. Changes in clinical symptoms of gallbladder polyps, use Visual Analogue Scale (VAS) to evaluate this indicator on weeks 12±1 and weeks 24±1.
3. Clinical safety indexes, use laboratory examination such as blood biochemical examination, routine blood test for safety observation on weeks 12±1 and weeks 24±1. Besides, observe and record the occurrence of adverse events (AE) of subjects from baseline to follow-up cycle finished.

ELIGIBILITY:
Inclusion Criteria:

Participants suitable for enrollment in this study must meet all of the following criteria:

1. Be between 18 and 75 years of age, male or female.
2. More than or equal to 2 gallbladder polyps were detected by B-ultrasound within 2 weeks before enrollment, and the maximum diameter of gallbladder polyps is between 3-7 mm.
3. No symptoms, or only some non-specific symptoms, such as ventosity, nausea, anorexia, right upper abdominal pain and right shoulder pain, etc.
4. Provide written informed consent.

Exclusion Criteria:

Participants who meet any of the following criteria will not be eligible for inclusion in this study:

1. Thickness of gallbladder wall is larger than 6 mm.
2. Clinically diagnosed as gallbladder cancer.
3. Clinically diagnosed as gallbladder and/or bile duct stones, and/or acute cholecystitis.
4. Previously performed gallbladder/biliary tract related operations, such as gallbladder-protected lithotomy, ERCP lithotomy, PTCS lithotomy and PTGBD.
5. Have severe infectious or severe primary diseases such as diseases in cardiovascular, cerebrovascular, pulmonary, renal or endocrine or hematopoietic system, or with mental diseases and/or behavioral abnormalities, which cannot be enrolled in the study determined by investigator.
6. Have irregular stool, and/or daily stool frequency more than or equal to 5 times in recent 2 weeks.
7. Regularly taken any Chinese patent medicine (including traditional Chinese medicine injection) with "soothing liver, cholagogic, clearing heat, dredging intestines" clearly written in the instructions, or regularly taken the traditional Chinese medicine decoction with the effect of soothing liver and cholagogic in recent 4 weeks.
8. Regularly taken proton pump inhibitors or H2 receptor antagonists or cholinergic receptor antagonists or gastrin receptor antagonists in recent 4 weeks.
9. Allergic to Danning Tablet and its components, has history of allergy, or has allergic constitution, or in allergic state.
10. Are pregnant, planning to be pregnant or breastfeeding.
11. Poor compliance, unable to cooperate with the investigator;
12. Have previously been involved in another clinical trial in the past three month;
13. Other situations not suitable for inclusion.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 336 (Estimated)
Dates: Start 2023-01-01 (Estimated); Primary Completion 2024-08-31 (Estimated); Study Completion 2024-11-30 (Estimated)

PRIMARY OUTCOMES:
Maximum diameter of gallbladder polyps on weeks 12±1 | weeks 12±1
  Use gallbladder ultrasonography to evaluate the maximum diameter of gallbladder polyps.
Maximum diameter of gallbladder polyps on weeks 24±1 | weeks 24±1
  Use gallbladder ultrasonography to evaluate the maximum diameter of gallbladder polyps.

SECONDARY OUTCOMES:
Thickness of gallbladder wall on weeks 12±1 | weeks 12±1
  Use gallbladder ultrasonography to evaluate thickness of gallbladder wall.
Thickness of gallbladder wall on weeks 24±1 | weeks 24±1
  Use gallbladder ultrasonography to evaluate thickness of gallbladder wall.
Level of abdominal pain on weeks 4±1 | weeks 4±1
  Use Visual Analogue Scale (VAS) to evaluate the level of abdominal pain caused by gallbladder polyps.
Level of abdominal pain on weeks 8±1 | weeks 8±1
  Use Visual Analogue Scale (VAS) to evaluate the level of abdominal pain caused by gallbladder polyps.
Level of abdominal pain on weeks 12±1 | weeks 12±1
  Use Visual Analogue Scale (VAS) to evaluate the level of abdominal pain caused by gallbladder polyps.
Level of abdominal pain on weeks 24±1 | weeks 24±1
  Use Visual Analogue Scale (VAS) to evaluate the level of abdominal pain caused by gallbladder polyps.
Clinical safety indexes | up to weeks 24±1
  Observe and record the occurrence of adverse events (AE) of subjects from baseline to follow-up cycle finished.

CONTACTS AND LOCATIONS:
Overall Officials: Feng Shen, MD, PhD, Principal Investigator — Eastern Hepatobiliary Surgery Hospital, Naval Medical University; Tian Yang, MD, PhD, Principal Investigator — Eastern Hepatobiliary Surgery Hospital, Naval Medical University
Locations (18):
- China (18):
  - The Second Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Xiangya Changde Hospital, Changde, Hunan
  - The First Affiliated Hospital of University of South China, Hengyang, Hunan
  - Loudi Central Hospital, Loudi, Hunan
  - Yiyang Central Hospital, Yiyang, Hunan
  - Affiliated Hospital of Nantong University, Nantong, Jiangsu
  - First Affiliated Hospital of Gannan Medical University, Ganzhou, Jiangxi
  - Shangrao People's Hospital, Shangrao, Jiangxi
  - Central Hospital Affiliated to Shandong First Medical University (Jinan Central Hospital), Jinan, Shandong
  - Shandong Provincial Third Hospital, Jinan, Shandong
  - The Affiliated Hospital of Qingdao University, Qingdao, Shandong
  - Eastern Hepatobiliary Surgery Hospital, Naval Medical University,, Shanghai, Shanghai Municipality
  - Shanxi Provincial People's Hospital, Taiyuan, Shanxi
  - The Sixth People's Hospital of Chengdu, Chengdu, Sichuan
  - Anning First People's Hospital, Anning, Yunan
  - Jinhua Municipal Central Hospital, Jinhua, Zhejiang
  - Ningbo Municipal Hospital of Traditional Chinese Medicine, Ningbo, Zhejiang
  - Affiliated Hospital of Shaoxing University, Shaoxing, Zhejiang